CLINICAL TRIAL: NCT01610297
Title: A Phase II, Multi-center, Single-arm, Prospective Study to Evaluate the Safety and Efficacy of Deferasirox in Beta-thalassemia Major Patients After Hematopoietic Stem Cell Transplantation.
Brief Title: Post Hematopoietic Stem Cell Transplantation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CICL670ATR04
Record Dates: First submitted 2012-05-30; First posted 2012-06-04 (Estimated); Results first posted 2016-07-21 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-09

CONDITIONS: Iron Overload After Hematopoietic Stem Cell Transplantation (HSCT) in Patients With Beta-thalassemia Major
Keywords: hematopoietic stem cell transplantation, beta-thalassemia major, deferasirox, iron overload
MeSH Terms: conditions — beta-Thalassemia; Iron Overload | interventions — Deferasirox

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ICL670 (Experimental): Oral dose of ICL670 at 10 mg/kg daily
  Interventions: Drug: ICL670

INTERVENTIONS:
Drug: ICL670 — Oral dose of ICL670 at 10 mg/kg daily

SUMMARY:
This was a prospective, single-arm, multicenter, national, phase II clinical study. The purpose of this Phase II study was to examine the safety and efficacy of deferasirox to decrease iron overload (IOL) in the posttransplant period in patients with beta-thalassemia major.

ELIGIBILITY:
Inclusion Criteria

* Patients who had hematopoietic stem cell transplantation (HSCT) for beta-thalassemia major
* hematopoietic stem cell transplantation (HSCT) was performed minimum 6 months and maximum 2 years ago
* The washout period after the immunosuppressive therapy should be at least 3 months.
* Signifacant IOL should be present including:

A. Serum ferritin >1000 μg/L or B. cardiac MRI <20 ms or C. liver iron concentration ≥ 5 mg/g dry weight measured by R2* MRI

Exclusion Criteria

* Patients who had any contraindication for treatment with deferasirox according to the prescribing information

  •Patients who depended on transfusion
* Patients with clinical symptoms of cardiac dysfunction (shortness of breath at rest or exertion, orthopnea, exercise intolerance, lower extremity edema, arrhythmias)
* Patients who were experiencing severe complication of HSCT e.g. acute Graft-versus host disease (GVHD)
* Significant proteinuria / Increase in serum creatinine

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2013-09; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- Turkey (Türkiye) (4):
  - Novartis Investigative Site, Ankara, Turkey
  - Novartis Investigative Site, Izmir, Turkey
  - Novartis Investigative Site, Antalya
  - Novartis Investigative Site, Istanbul

REFERENCES:
- [Derived] Yesilipek MA, Karasu G, Kaya Z, Kuskonmaz BB, Uygun V, Dag I, Ozudogru O, Ertem M. A Phase II, Multicenter, Single-Arm Study to Evaluate the Safety and Efficacy of Deferasirox after Hematopoietic Stem Cell Transplantation in Children with beta-Thalassemia Major. Biol Blood Marrow Transplant. 2018 Mar;24(3):613-618. doi: 10.1016/j.bbmt.2017.11.006. Epub 2017 Nov 16. PMID 29155313

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ICL670
Started | 27
Completed | 26
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | ICL670
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.07 (3.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events, Serious Adverse Events and Deaths as a Measure of Safety and Tolerability
Description: To determine the safety; incidence, type and severity of adverse events including renal, hepatic, biochemistry and hematologic parameters of deferasirox in the treatment of iron overload after hematopoietic stem cell transplantation (HSCT) in patients with beta-thalassemia major in 12 months period
Time Frame: 12 months
Population: The Safety Set (SS) includes all included patients who were included in the study. All statistical analyses of safety and tolerability will be done in the SS.
Measure: Number; unit: Participants
Arm/Group | ICL670
Number analyzed (Participants) | 27
Participants
  Adverse events | 25
  Serious adverse events | 3
  Death | 0

2. Secondary Outcome: Change in Serum Ferritin Level.
Description: Blood samples were collected and serum levels were assessed at study baseline (BL) and at 12 months.
Time Frame: Baseline, 12 Months
Population: The Full Analysis Set (FAS) comprises all patients in whom study treatment has been started and received at least one dose.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ICL670
Number analyzed (Participants) | 27
ng/mL
  Baseline | 1766.81 (599.64)
  Month 12 | 903.56 (596.62)

3. Secondary Outcome: Change in the Further Parameters of Iron Overload (Liver Iron Concentration by Magnetic Resonance Imaging (MRI Examination)
Description: Liver Iron Concentration (LIC) values between 3 and 7 mg Fe / g dry weight are indicative of mild iron deposition, while values between 7 and 15 mg Fe / g dry weight are indicative of moderate iron deposition which have been associated with liver disease. Values >15 mg Fe/g dry weight are indicative of severe iron deposition which is associated with progressive liver fibrosis, increased morbidity and mortality
Time Frame: Baseline, 12 month
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg Fe/g dry liver weight
Arm/Group | ICL670
Number analyzed (Participants) | 27
mg Fe/g dry liver weight
  Baseline Liver MRI(n= 27) | 12.07 (9.42)
  Week 52 Liver MRI (n=25) | 4.62 (2.85)

4. Secondary Outcome: The Percentage of Patients Reaching Serum Ferritin Levels Lower Than 500 μg/L
Description: Serum Ferritin values between 1000-2500 μg/L are indicative of mild to moderate iron overload while values >2500 μg/L are indicative of severe iron overload and levels constantly higher than 2500 μg/L has been shown to to increase the risk of cardiac complications and endocrine disease. Maintaining levels <1000 μg/L is associated with increased survival and less morbidity.
Time Frame: Week 28 and Week 52
Population: as for outcome 2
Measure: Number; unit: Percentage of Patients
Arm/Group | ICL670
Number analyzed (Participants) | 27
Percentage of Patients
  Week 28 (n=26) | 7.7
  Week 52 (n=27) | 33.3

5. Secondary Outcome: Change in the Further Parameters of Iron Overload (Cardiac Iron Concentration by Magnetic Resonance Imaging (MRI Examination)
Description: Cardiac MRI values between 10 to 20 milliseconds (ms) are indicative of moderate cardiac iron deposition associated with declining left ventricular ejection fraction and arrhythmias while values <10 ms are indicative of deposition sufficient to risk cardiac decompensation and associated with overt heart failure and mortality.
Time Frame: Baseline, 12 month
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | ICL670
Number analyzed (Participants) | 27
ms
  Baseline Cardiac MRI(n= 27) | 26.48 (7.49)
  Week 52 Cardiac MRI (n=24) | 28.25 (5.53)

ADVERSE EVENTS:
Arm/Group | ICL670
Serious Adverse Events (participants affected / at risk) | 3/27
Other Adverse Events (participants affected / at risk) | 23/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ICL670 (N=27)
Neutrophil count decreased (Investigations) | 2
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Influenza like illness (General disorders) | 1
Office visit (Surgical and medical procedures) | 1
Hepatitis B (Hepatobiliary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ICL670 (N=27)
Anemia (Blood and lymphatic system disorders) | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Pyrexia (General disorders) | 7
Aspartate aminotransferase increased (Investigations) | 6
Pharyngitis (Infections and infestations) | 6
Influenza (Respiratory, thoracic and mediastinal disorders) | 5
Diarrhea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 3
White blood cell count decreased (Investigations) | 2
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 2
Eczema (Skin and subcutaneous tissue disorders) | 2
Haemophilus infection (Infections and infestations) | 2
Herpes zoster (Infections and infestations) | 2
Hypersensitivity (Immune system disorders) | 2
Infection (Infections and infestations) | 2
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 2
Sinusitis (Infections and infestations) | 2
Alanine aminotransferase increased (Investigations) | 7
Influenza like illness (General disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.